CLINICAL TRIAL: NCT00874419
Title: A Randomized, Open-label, Multi-center Phase III Study of Erlotinib Versus Gemcitabine/Carboplatin in Chemo-naive Stage IIIB/IV Non-Small Cell Lung Cancer Patients With EGFR Exon 19 or 21 Mutation (Optimal)
Brief Title: Erlotinib Versus Gemcitabine/Carboplatin in Chemo-naive Stage IIIB/IV Non-Small Cell Lung Cancer Patients With Epidermal Growth Factor Receptor (EGFR) Exon 19 or 21 Mutation
Acronym: ML20981
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tongji University (Other)
Collaborators: Sun Yat-sen University (Other); Shanghai Chest Hospital (Other); RenJi Hospital (Other); Guangdong Provincial People's Hospital (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Shanghai Pulmonary Hospital, Tongji University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20981
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: EGFR mutation; EGFR-TKI; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- erlotinib (Experimental): Arm 1 receive erlotinib 150 mg oral, once a day until progression or unacceptable toxicity
  Interventions: Drug: erlotinib
- gemcitabine/carboplatin (Active Comparator): gemcitabine 1000mg/m2 on d1,8 with carboplatin AUC=5 on d1 intravenously, every 3 weeks, up to 4 cycles
  Interventions: Drug: gemcitabine/carboplatin

INTERVENTIONS:
Drug: erlotinib — erlotinib 150 mg oral, once a day
  Other Names: Tarceva
  Arms: erlotinib
Drug: gemcitabine/carboplatin — gemcitabine 1000mg/m2 on d1,8 with carboplatin AUC=5 on d1 intravenously, every 3 weeks, up to 4 cycles
  Other Names: Gemzar
  Arms: gemcitabine/carboplatin

SUMMARY:
Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR TKIs) such as erlotinib have proved effective in second or third line therapy for advanced non-small cell lung cancer(NSCLC).It is well tolerated without the side effects usually associated with chemotherapy. The mutations in EGFR exons 19 or 21 have been reported to be associated with efficacy of EGFR TKIs.Based on the encouraging preliminary results from the Spanish lung cancer group' prospective study reported that the efficacy of Tarceva as first line treatment for metastatic NSCLC patients with EGFR mutation would delay disease progression,prolong overall survival and be well tolerated, medium Progression-free survival(PFS) was around 12 months and OS reach 24 months，our study is designed to compare PFS between the patients with mutant EGFR treated by gemcitabine/carboplatin and those by erlotinib in the first-line setting. We assumed 11 months of PFS on Tarceva arm versus 6 months on chemotherapy arm with a=0.025(alpha-spend for an interim analysis), 80% power and 12 months enrolment period, 12 months FU duration to calculate the sample size. The sample size is 69 pairs. Considering about 10% drop-out rate, the final sample size is 152 patients.So, chemo-naive staged IIIb/IV patients with EGFR mutations in exon 19 or 21 will be enrolled into this open-label, randomized,multicenter phase III study.

DETAILED DESCRIPTION:
Primary Outcome Measures:

Progression-free survival(PFS) Secondary Outcome Measures: Overall response rate(ORR), overall survival(OS), quality of life(QOL),etc.

Estimated Enrollment: 160 Study Start Date: August 2008 Estimated Study Completion Date: August 2010

The patients will be randomized into the following two arms:

Arm A: erlotinib 150mg once per day up to disease progression or intolerable toxicity.

Arm B: Gemcitabine (1000mg/m2, IV,d1 and d8) plus Carboplatin (AUC=5, IV d1) repeated every 3 weeks up to 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IIIB (cytological confirmed with malignant pleural effusion or pericardial effusion) or histopathological or cytological confirmed stage IV NSCLC or relapsed after complete resection .
2. EGFR exon19 deletions or exon 21 L858R mutation by the DNA direct PCR sequencing using fresh tumor sample or paraffin embed tumor sample.
3. Measurable lesions as defined by RECIST criteria .
4. Palliative radiotherapy allowed if it was finished 3 weeks after the first drug administration, but the target lesions should not be included in the radiotherapy field.
5. Patients with operation are allowed if the operation is 4 weeks before the first drug administration
6. Men or women of at least 18 years of age.
7. ECOG Performance status of 0 to 2.
8. Estimated life expectancy of at least 12 weeks.
9. Patient compliance and geographic proximity that allow adequate follow-up.
10. Adequate organ function tested 7 days before the first drug administration:

    hemoglobin ≥9 g/dL,absolute neutrophil count (ANC) ≥1.5*109/L, platelets ≥100 *109/L,bilirubin ≤1.5ULN, alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 upper limited number(ULN) (AP, AST, ALT ≤5ULN is acceptable if liver has tumor involvement).INR≤1.5, APTT in the normal range( 1.2DLN-1.2ULN),creatinine ≤1.5ULN.
11. Informed consent from the patient.

Exclusion Criteria:

1. Have received systemic anti-cancer therapy, including Cytotoxic drugs, targeted therapy, experimental treatment, adjuvant or neo-adjuvant therapy(except the disease relapse 6 months after the final drug)
2. Wild type EGFR.
3. Uncontrolled pericardial or pleural effusions prior to study entry.
4. History of cardiovascular disease: Congestive Heart Failure > grade II in NYHA. Unstable angina patients (have angina symptoms in rest) or a new occurrence of angina (began in the last 3 months) or myocardial infarction happens in the last 6 months
5. Brain metastasis (controlled brain metastasis and steroid free need is excluded).
6. HIV infection
7. Active infection, >grade 2 in Common Terminology Criteria for Adverse Events(CTCAE) version 3.
8. A history of operation or serious traumatic 3 weeks before the first drug administration
9. Patient with other malignant tumor except NSCLC 5 years previous to study entry. Excluding cervical carcinoma in situ, cured basal cell carcinoma, bladder epithelial tumor [including Ta and Tis]
10. Mixed with small cell lung cancer
11. Unable to swallow drugs.
12. Malabsorption
13. Pregnant or child breast feeding women
14. Childbearing patients will not use a reliable method of contraception before the study entry, during process of the study and within 30 days after discontinuation of the study. Reliable contraceptive methods will be determined by principal investigator or a designated officer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 12 months

SECONDARY OUTCOMES:
OS | 24 months
ORR | 24 months
Time to Progression | 24 months
lung cancer symptoms and health-related quality of life (HRQoL) | 24 months
explore the biological markers (tumor tissue) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD & PhD, Principal Investigator — Tongji University
Locations (1):
- Medical Department, Shanghai Pulmonary Hospital, Shanghai, China

REFERENCES:
- [Derived] Zhou C, Wu YL, Chen G, Feng J, Liu XQ, Wang C, Zhang S, Wang J, Zhou S, Ren S, Lu S, Zhang L, Hu C, Hu C, Luo Y, Chen L, Ye M, Huang J, Zhi X, Zhang Y, Xiu Q, Ma J, Zhang L, You C. Final overall survival results from a randomised, phase III study of erlotinib versus chemotherapy as first-line treatment of EGFR mutation-positive advanced non-small-cell lung cancer (OPTIMAL, CTONG-0802). Ann Oncol. 2015 Sep;26(9):1877-1883. doi: 10.1093/annonc/mdv276. Epub 2015 Jul 3. PMID 26141208
- [Derived] Zhou C, Wu YL, Chen G, Feng J, Liu XQ, Wang C, Zhang S, Wang J, Zhou S, Ren S, Lu S, Zhang L, Hu C, Hu C, Luo Y, Chen L, Ye M, Huang J, Zhi X, Zhang Y, Xiu Q, Ma J, Zhang L, You C. Erlotinib versus chemotherapy as first-line treatment for patients with advanced EGFR mutation-positive non-small-cell lung cancer (OPTIMAL, CTONG-0802): a multicentre, open-label, randomised, phase 3 study. Lancet Oncol. 2011 Aug;12(8):735-42. doi: 10.1016/S1470-2045(11)70184-X. Epub 2011 Jul 23. PMID 21783417